CLINICAL TRIAL: NCT00478465
Title: A Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Efficacy and Safety of Valganciclovir (Valcyte) in Patients Experiencing Chronic Fatigue Syndrome With Elevated Antibody Titers Against Human Herpesvirus-6 (HHV-6) and Epstein-Barr Virus (EBV)
Brief Title: Valganciclovir (Valcyte) for Chronic Fatigue Syndrome Patients Who Have Elevated Antibody Titers Against Human Herpes Virus 6 (HHV-6)and Epstein-Barr Virus (EBV)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MV21103 Version 3.0
Record Dates: First submitted 2007-05-23; First posted 2007-05-24 (Estimated); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Chronic Fatigue Syndrome
Keywords: chronic fatigue syndrome; fatigue; valganciclovir; valcyte; Epstein-Barr virus; EBV; Human herpes virus 6; HHV 6; herpes viruses; herpes
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Fatigue; Epstein-Barr Virus Infections; Herpes Simplex | interventions — Valganciclovir

INTERVENTIONS:
Drug: valganciclovir

SUMMARY:
The purpose of this study determine whether the drug valganciclovir has a significant and real benefit on the central core of symptoms experienced by patients who have high titers to EBV and HHV-6 and are experiencing long-standing fatigue and cognitive impairment (CFS).

In addition, to characterize a quantifiable biological marker in these patients that will facilitate the identification of those likely to respond to valganciclovir and will make it possible to assess response to treatment.

DETAILED DESCRIPTION:
Chronic fatigue syndrome (CFS) is a clinically defined condition characterized by severe disabling fatigue and a combination of symptoms that prominently features self-reported impairment of concentration and short-term memory, sleep disturbances, and musculoskeletal pain. Prevalence of CFS in the adult population is estimated to be 0.007% to 2.8%. No pathognomonic signs or diagnostic tests for this condition have been yet validated in scientific studies; in addition, no definitive treatments are clinically available. Suggested etiologies of CFS include, but are not limited to: viral or bacterial infections, endocrine-metabolic dysfunction, immunological imbalance, neurally-mediated hypotension and depressioN. EBV and HHV-6 are among the viruses frequently thought as associated with CFS.

We recently encountered a group of patients at Stanford who were chronically infected with human herpes virus 6 (HHV-6) and Epstein-Barr virus (EBV), were suffering from debilitating fatigue for at least one year and experienced a significant improvement in their fatigue and cognitive symptoms following the administration of valganciclovir. Their antibody titers to both viruses were high (median antibody titer for EBV viral capsid antigen was 1:2560 and for HHV-6 IgG was 1:1280) despite the fact that some of them were known to have been infected with EBV and HHV-6 for several years. We suspected that their symptoms could be the result of an immune dysregulation triggered by high levels of replication of both EBV and HHV-6 (alterations in the immune system such as an aberrant cytokine profiles have been proposed as the central abnormality in patients with CFS associated with other viruses such as parvovirus B19. At the same time, we were familiar using valganciclovir in the context of several clinical settings including its known indications for reactivation of viral infections in immunocompromised patients. We were comfortable using valganciclovir (900 mg bid for three weeks followed by 900 mg qd to complete 3 to 12 months of treatment) in patients with solid and bone marrow transplants, cancer or other immunosuppressive disorders who had developed CMV, EBV, or HHV-6 disease.

We hypothesized that a long course (i.e. 6 months) of valganciclovir could effectively decrease or stop ongoing viral replication of both EBV and HHV-6 and that this virological effect could be translated in a clinical and laboratory benefit (i.e. decrease or resolution of lymphadenopathy, reversion of the CD4/CD8 ratio abnormalities). We were surprised to see that a dramatic recovery on the level of physical activity was also observed in the Stanford patients (from a median of 10% of energy level for daily activities at baseline to 90% after valganciclovir use). Of note, the drug has also been tried in patients in whom an improvement on their level of physical activity has not been observed. The total number of patients treated today is 30, 26 had "elevated titers" and 4 had "low titers". Of the 26 patients with "elevated titers", 25 have had a dramatic recovery. Of the 4 patients with "low titers", none have responded.

We believe that our successful experience with valganciclovir in a subset of patients with CFS at Stanford calls for a prospective study to exclude a placebo effect. We propose to measure viral, immunologic, and genomic endpoints to assess whether there are objective and measurable changes in these parameters and whether they correlate with clinical improvement. Clinical improvement will be assessed by objective measurements of daily physical and psychological activities. This will help to elucidate the possible role of HHV-6, EBV (or a yet to be known virus) and/or an altered immune system as triggers for the symptoms experienced by patients suffering CFS and to establish whether the drug valganciclovir does reverse these abnormalities. This study may also shed light on a biomarker or profile of biomarkers associated with (or diagnostic of) CFS.

We will be executing a randomized, double-blind, placebo-controlled clinical trial to evaluate the efficacy and safety of valganciclovir in patients experiencing chronic fatigue syndrome with elevated antibody titres against Human Herpesvirus-6 (HHV-6) and Epstein-Barr Virus (EBV)

Objectives

1. To determine whether the drug valganciclovir has a significant and real benefit on the central core of symptoms experienced by patients who have high titers to EBV and HHV-6 and are experiencing long-standing fatigue and cognitive impairment (CFS).
2. To characterize a quantifiable biological marker in these patients that will facilitate the identification of those likely to respond to valganciclovir and will make it possible to assess response to treatment.

Design of the study A double-blind, placebo-controlled, randomized clinical trial. All patients will be given the active drug (20 patients) or placebo (10 patients) for 6 months and followed for an additional 3 months. Patients on the placebo arm will take a valganciclovir look-alike tablet that does not contain the active drug for the initial six month period. Subsequently these patients will be offered a 6 month trial of valganciclovir if at the end of the study (when the last enrolled patient reaches 9 months from initiating therapy) it is clear that there is a benefit of valganciclovir therapy and patients have not spontaneously improved.

Kogelnik A, Rosso F, Hoegh-Petersen M and Montoya JG. Use of Valganciclovir in Patients Chronically Co-infected with Human Herpes Virus 6 (HHV-6) and Epstein-Barr Virus (EBV) who were Experiencing Long-standing Fatigue. J Clin Virol 2006 Volume 37, Supplement 1 S33-S38

Kerr JR, Cunniffe VS, Kelleher P, Bernstein RM and Bruce IN. Successful intravenous immunoglobulin therapy in 3 cases of parvovirus B19-associated chronic fatigue syndrome. Clin Infect Dis 2003;36:e100-6

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥ 18 years old).
2. Patient understands and signs the Informed Consent.
3. Patients who meet the clinical criteria for the diagnosis of chronic fatigue syndrome as established by the International Chronic Fatigue Syndrome Study Group in 1994 [10].
4. Patients who had a "viral onset" for their CFS.
5. Patients whose CFS symptoms are not spontaneously improving and have plateau for at least 6 months.
6. Patients with "high" antibody titers against HHV-6 IgG ≥ 640, EBV VCA IgG ≥ 640 and detectable EA Ab at 1:160 or HHV-6 IgG ≥ 320 if EBV VCA IgG ≥ 1280 and has detectable EA Ab at 1:160 (measured by the average of a minimum of two time points obtained during screening at least 3 weeks apart).
7. Patient agrees to utilize two reliable methods of contraception combined throughout the study period and for 90 days following discontinuation of the Study Drug.
8. Females of childbearing potential will have a negative pregnancy test at screening.

Exclusion Criteria:

1. Patients who are found to have alternate medical and/or psychiatric causes for their fatigue (see guidelines established by the International Chronic Fatigue Syndrome Study Group in 1994 [1].
2. Patients with history of major depression with psychotic or melancholic features before the diagnosis of CFS or who are found to be actively depressed (major depression with psychotic or melancholic features) by the depression instrument used for the study and by a medical evaluation by a psychiatrist.
3. Patients with other serious co-morbidities which according to the investigator may interfere with the ability of the patient to participate in the study
4. Patients with history of substance abuse in the past year (excluding nicotine and caffeine) or positive urine test for substance abuse.
5. Patients with any other known chronic viral orbacterial infection for which other treatment(s) is(are) available
6. Patients with an active concurrent acute infection
7. Patients with abnormal creatinine clearance (≤60ml/min)
8. Patients with ANC ≤1500 /mm3
9. Patients with Hb ≤ 10 g/dl
10. Patients with platelet count ≤ 100 000/mm3
11. Previous hypersensitivity or contraindication to Valganciclovir/ganciclovir
12. Patients taking other antiviral medications or who have received antiviral medications within the previous three months
13. Patients receiving other experimental therapy
14. Patient is simultaneously participating in another clinical trial
15. Patient requires the use of any prohibited concomitant medications (see Insert on VALCYTE prescribing information).
16. Women in childbearing age considering getting pregnant during the study period
17. Patient is a lactating female who will not discontinue nursing prior to study entry. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-05 (Actual); Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose G Montoya, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Medical Center, Stanford, California, United States

REFERENCES:
- [Derived] Montoya JG, Kogelnik AM, Bhangoo M, Lunn MR, Flamand L, Merrihew LE, Watt T, Kubo JT, Paik J, Desai M. Randomized clinical trial to evaluate the efficacy and safety of valganciclovir in a subset of patients with chronic fatigue syndrome. J Med Virol. 2013 Dec;85(12):2101-9. doi: 10.1002/jmv.23713. Epub 2013 Aug 19. PMID 23959519